CLINICAL TRIAL: NCT05675865
Title: Cryoablation for Monomorphic Ventricular Tachycardia IDE Study: EFS and Pivotal
Brief Title: Cryoablation for Monomorphic Ventricular Tachycardia
Acronym: FULCRUM-VT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Adagio Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CS-300
Record Dates: First submitted 2022-12-14; First posted 2023-01-09 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Sustained VT
Keywords: cryoablation; monomorphic VT; sustained monomorphic VT

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- VT Cryoablation (Experimental): all enrolled patients will have a ablation procedure using the Adagio VT Cryoablation System for SMVT
  Interventions: Device: cryoablation procedure

INTERVENTIONS:
Device: cryoablation procedure — ablation procedure for VT using the investigational device

SUMMARY:
The objective of this clinical study is to evaluate the safety and effectiveness of the Adagio VT Cryoablation System in the ablation treatment of Sustained Monomorphic Ventricular Tachycardia (SMVT)

DETAILED DESCRIPTION:
A prospective, single-arm, multi-center, open label, pre-market, clinical study designed to provide safety and efficacy data regarding the use of the Adagio System in the treatment of scar-mediated SMVT in ischemic and non-ischemic patients.

Study subjects will include patients who experience recurrent SMVT and are scheduled for an endocardial VT ablation.

Study subjects must have an Implantable Cardioverter Defibrillator (ICD) prior to the cryoablation procedure.

This IDE study includes two phases, an early feasibility (EFS) phase to support initial device safety and effectiveness, and a Pivotal Study phase to collect safety and effectiveness data for a future PMA marketing application.

ELIGIBILITY:
Inclusion Criteria (IC):

* IC 1 Male or female ≥ 18 years
* IC 2 Patients with a clinical indication for catheter ablation due to ischemic and/or non-ischemic heart disease and recurrent symptomatic sustained scar-mediated monomorphic Ventricular Tachycardia.
* IC 3 Any of the following:

  * Ischemic cardiomyopapthy (ICM) patients with prior history of myocardial infarction with Q waves, focal wall motion abnormality on imaging, fixed perfusion defect correlating with coronary stenosis or prior coronary intervention, 20% ≤ LVEF < 50%.
  * non-ischemic cardiomyopathy (NICM) patients with scar in a territory without coronary stenosis as evidenced by CMR imaging within the prior 90 days or intra-procedurally using EAM and PES prior to investigational device use, 20% ≤ LVEF < 50%
  * Arrhythmogenic right ventricular cardiomyopathy (ARVC)
* IC 4 Has received a market-released ICD prior to enrollment
* IC 5 Patient has had at least 1 documented spontaneous episode of SMVT within the previous 6 months
* IC 6 Refractory to, or intolerant of, at least one Class III AAD. (Refractory or intolerant defined as AAD failure due to recurrent VT, not tolerated/ desired due to side effects)
* IC 7 Willingness, ability, and commitment to participate in baseline and follow-up evaluations for the full length of the study
* IC 8 Willingness and ability to give an informed consent

Exclusion Criteria (EC):

* EC 1 Intracardiac thrombus by TTE or TEE within 48 hours prior to the procedure
* EC 2 Presence of isolated epicardial scar(s) requiring epicardial ablation identified by either preoperative CMR imaging within 90 days of procedure or intra-procedurally using EAM and PES prior to investigational device use
* EC 3 VTs due to any of the following causes:

  1. Idiopathic VT
  2. Automaticity or triggered activity
  3. Bundle Branch Reentry (BBR)
  4. Any focal tachycardia (e.g., papillary, RVOT)
  5. Ventricular tachycardia secondary to electrolyte imbalance, active thyroid disease, or any other reversible or non-cardiac cause
* EC 4 NICM patients only, if any of the following apply:

  1. Congenital condition that limits access to the left or right ventricles
  2. Severe aortic or mitral stenosis, severe mitral regurgitation, or severe aortic insufficiency
  3. Active inflammatory processes (e.g., myocarditis) within the past 120 days
  4. Sarcoidosis
  5. Hypertrophic cardiomyopathy
  6. Drug- or alcohol-induced cardiomyopathy
* EC 5 Any VT ablation within 4 weeks prior to enrollment
* EC 6 More than one prior (>4 weeks) VT ablation or prior surgical treatment for VT within the past 2 years
* EC 7 Cardiogenic shock, unless it is due to incessant monomorphic VT
* EC 8 Any other cardiovascular conditions as described below:

  1. Class IV heart failure
  2. Aortic aneurysm
  3. Previous cardiac surgery or percutaneous coronary intervention within 60 days prior to index procedure
  4. Interatrial baffle, closure device, patch, or PFO occlusion device
  5. Coronary artery bypass graft (CABG) procedure within six (6) months prior to the ablation procedure
  6. Acute MI or unstable angina in the previous 60 days
  7. Mechanical mitral or aortic valve
  8. Cardiac myxoma
  9. Significant congenital heart disease
* EC 9 Acute illness or active systemic infection
* EC 10 Any previous history of cryoglobulinemia
* EC 11 History of blood clotting or bleeding disease
* EC 12 Peripheral vascular disease that precludes LV access
* EC 13 Contraindication to heparin
* EC 14 Allergy to radiographic contrast dye that cannot be medically managed prior to the ablation procedure
* EC 15 Any prior history of documented cerebral vascular accident (CVA), TIA or systemic embolism (excluding a post-operative Deep Vein Thrombosis, DVT), within 6 months prior to the ablation procedure.
* EC 16 Pregnant, or anticipated pregnancy during study follow-up
* EC 17 Current enrollment in any other study protocol where testing or results from that study may interfere with the procedure or outcome measurements for this study
* EC 18 Any other condition (e.g., ARVC with extensive free wall scarring) that, in the judgment of the investigator, makes the patient a poor candidate for this procedure, the study or compliance with the protocol (includes vulnerable patient population, mental illness, addictive disease, candidate for heart transplantation, patient with ventricular assist device, or terminal illness with a life expectancy less than 12 months)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Estimated)
Dates: Start 2023-09-11 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Primary Safety Endpoint for EFS and Pivotal phases is freedom from definite or probable device or procedure related Major Adverse Events (MAEs) that occur within 7 days following the cryoablation procedure. | 7 days following the ablation procedure
  Events will be adjudicated by an independent Clinical Events Committee (CEC). MAEs include any of the following:
  * Death
  * Acute myocardial infarction
  * Cardiac perforation/pericardial tamponade
  * Cerebral infarct or systemic embolism
  * Major bleeding requiring transfusion
  * Acute Mitral, Tricuspid or Aortic valve damage resulting in moderate or severe regurgitation
  * Access site complications requiring medical or surgical intervention
  * Pericarditis
  * Heart block requiring a permanent pacemaker
  * Other serious adverse device effects (SADEs), including TIAs, adjudicated by an independent Clinical Events Committee (CEC) to be probably or definitely related to the Adagio System.
Primary Procedural Endpoint for EFS and Pivotal - Analysis of the proportion of subjects with non-inducible VT or no further ablation targets meeting the criteria for ablation at the end of the cryoablation procedure. | During Procedure
  Documentation of non-inducibility of any VT targeted for ablation at the end of procedure.
Primary Efficacy Endpoint for Pivotal Phase | 6 months after the procedure
  Defined as freedom from recurrent sustained MMVT in the absence of a new AAD or increase in dose of a pre-ablation AAD for VT management at 6 months following the ablation procedure, where sustained MMVT is defined as continuous MMVT for > 30 seconds (programmed monitoring zone only), or MMVT requiring appropriate ICD intervention regardless of duration. All ICD interrogation reports will be adjudicated by an independent VT Event Committee (VTEC) to support the primary efficacy endpoint.

SECONDARY OUTCOMES:
Secondary Safety Endpoint - Analysis of the proportion of subjects with freedom from definite or probable device or procedure related MAEs that occur within 30 days (EFS) or SAEs within 12 months (pivotal) following the cryoablation procedure. | 1 month post cryoablation procedure
  Events will be adjudicated by an independent Clinical Events Committee (CEC).
Secondary Efficacy Endpoint for EFS and Pivotal - Analysis of the proportion of subjects with freedom from inducible MMVT <30s | 6-month post cryoablation procedure
  Freedom from inducible MMVT with a cycle length similar to (within 30 ms) or slower than the targeted VT and lasting longer than 30 seconds at the end of the ablation procedure.
Secondary Efficacy Endpoint for EFS and Pivotal - Analysis of the proportion of subjects with freedom from VT > 30 seconds | 6-month post cryoablation procedure
  Freedom from Ventricular Tachycardia lasting longer than 30 seconds or appropriate ICD intervention at 6 months (EFS) or 12 months (pivotal).
Secondary Efficacy Endpoint for EFS and Pivotal - Analysis of the proportion of subjects with freedom from VT > 30 seconds without AAD | 6-month post cryoablation procedure
  Freedom from Ventricular Tachycardia lasting longer than 30 seconds or appropriate ICD intervention at 6 months in the absence of new AADs or increase in dose of pre-ablation AADs. Drug changes related specifically to management of atrial arrhythmias will not be included in the analysis of this endpoint (EFS
Health Outcomes for EFS and Pivotal phases are defined as all-cause mortality at 12 months | 12-months post cryoablation procedure
  All-cause mortality at 12 months
Health Outcomes for EFS and Pivotal phases are defined as cardiac mortality at 12 months | 12-months post cryoablation procedure
  Cardiac mortality at 12 months
Health Outcomes for EFS and Pivotal phases are defined as quality-of-life improvement as measured by reduction of VT burden at 6 and 12 months compared to baseline. | 6 and 12-months post cryoablation procedure
  Reduction in the number of ICD shocks and number of VT related hospitalizations

CONTACTS AND LOCATIONS:
Locations (15):
- United States (13):
  - Banner University Medical Center Phoenix, Phoenix, Arizona
  - University of California San Francisco, San Francisco, California
  - Johns Hopkins University, Baltimore, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Weill Cornell Medical Center, New York, New York
  - Northwell Health- Staten Island University Hospital, Staten Island, New York
  - Ohio State University, Columbus, Ohio
  - Hospital of University of Pennsylvania, Philadelphia, Pennsylvania
  - Medical Center of South Carolina (MUSC), Charleston, South Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Texas Cardiac Arrhythmia Research Institute (TCARF), Austin, Texas
- Canada (2):
  - Montreal Heart Institute, Montreal, Quebec
  - McGill University, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Weiss JP, Reddy VY, Tandri H, Richardson TD, Gerstenfeld EP, Stevenson WG, Jubran N, Grigorov I, Tung R. Ultra-Low Cryoablation for Scar-Related VT Ablation: Results From the US Early Feasibility Study. Circ Arrhythm Electrophysiol. 2026 Feb 2:e014095. doi: 10.1161/CIRCEP.125.014095. Online ahead of print. PMID 41623095